CLINICAL TRIAL: NCT00218972
Title: Physical Exercise in Hypertension, Randomised Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Traininghypertension; NCT00805363 (obsolete NCT alias)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: Hypertension
Keywords: Hypertension; endurance training; endothelial function; left ventricular function; Echocardiography; Quality of life; Essential hypertension grade 1 - 2
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- AIT: aerobic interval training (Active Comparator): High intensity interval training on treadmill at > 90% of maximal HR for four bouts of four minutes with warm up, active pauses and cool down, three times per week for 12 weeks.
  Interventions: Behavioral: Aerobic interval training
- MIT, moderate intensity training (Active Comparator): Moderate intensity treadmill continuous exercise at 70% of maximum heart rate for 47 minutes (in order to ensure isocaloric training amount), three times per week for 12 weeks.
  Interventions: Behavioral: moderate intensity training
- Recommendation of regular exercise (Active Comparator): No training intervention, general advice as prescribed in guidelines.
  Interventions: Behavioral: Recommendation of regular exercise

INTERVENTIONS:
Behavioral: Aerobic interval training
  Arms: AIT: aerobic interval training
Behavioral: moderate intensity training
  Arms: MIT, moderate intensity training
Behavioral: Recommendation of regular exercise
  Arms: Recommendation of regular exercise

SUMMARY:
Endurance training has a documented effect on hypertension. However, only low to moderate training intensity has so far been studied. High aerobic intensity should, from physiological considerations, prove more effective in also reducing high blood pressure. The present study is a randomised comparison of high versus moderate intensity versus training in groups, and general advice on 24 hour blood pressure in hypertensives. The training period is 12 weeks, with follow-up after 1 year. Maximum oxygen uptake, quality of life, left ventricular function and blood vessel reactivity are also measured.

DETAILED DESCRIPTION:
Endurance training has documented effect on blood pressure in hypertension. However, only low to moderate training intensity has so far been studied. Higher aerobic intensity based on individual measurements of maximum oxygen uptake is more efficient in increasing oxygen uptake, and might prove more effective in lowering blood pressure. Group training, on the other hand is not individualised, but less personnel required and may prove more cost effective. Endurance training is shown to improve both systolic and diastolic left ventricular function, as well as endothelial function. Both can be measured non-invasively by ultrasound.

The study is an open, randomised study with four arms, comparing:

* High aerobic intensity interval training
* Moderate aerobic intensity training
* Group training
* Controls receiving standard advice on lifestyle and training

Training effect is measured by Max. Oxygen uptake, blood pressure by continuous 24 hour ambulatory measurement, Left ventricular function by echo Doppler and endothelial function by flow mediated vasodilation by ultrasound.

The effect of exercise on blood pressure is dependent on continued training. All patients will be followed up after one year.

ELIGIBILITY:
Inclusion Criteria:

* Essential hypertension grade 1 - 2 without medical treatment

Exclusion Criteria:

* End organ damage
* Two or more cardiovascular risk factors
* Diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2005-02; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
24 hour blood pressure | 12 weeks

SECONDARY OUTCOMES:
Maximum oxygen uptake | 12 weeks
Endothelial function | 12 weeks
Echocardiographic left ventricular function | 12 weeks
Quality of life | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Asbjorn Stoylen, Dr. Med, Study Director — Dept. of Circulation and Medical Imaging, Faculty of Medicine, Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Result] Molmen-Hansen HE, Stolen T, Tjonna AE, Aamot IL, Ekeberg IS, Tyldum GA, Wisloff U, Ingul CB, Stoylen A. Aerobic interval training reduces blood pressure and improves myocardial function in hypertensive patients. Eur J Prev Cardiol. 2012 Apr;19(2):151-60. doi: 10.1177/1741826711400512. Epub 2011 Mar 4. PMID 21450580